CLINICAL TRIAL: NCT06557252
Title: The Application of the PDCA Management Model in Improving the Diagnostic Accuracy of AIG
Status: Not yet recruiting | Type: Observational
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-091A-01
Record Dates: First submitted 2024-08-12; First posted 2024-08-16 (Actual); Last update posted 2024-08-16 (Actual); Status verified 2024-08

CONDITIONS: Autoimmune Gastritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- not received PDCA training: no intervention
- PDCA training: The group of endoscopists underwent PDCA training to observe whether it ultimately improved the diagnosis rate of autoimmune gastritis.
  Interventions: Behavioral: PDCA training

INTERVENTIONS:
Behavioral: PDCA training — Improve diagnostic rate
  Groups: PDCA training

SUMMARY:
Autoimmune gastritis is currently relatively rare in China due to its insidious onset, diverse clinical manifestations involving multiple systems such as digestive, hematological, and nervous systems, and its association with other autoimmune diseases. It can also be complicated by hyperplastic gastric polyps, gastric neuroendocrine tumors, gastric adenocarcinoma, and other diseases, making it prone to clinical misdiagnosis. As a form of gastritis in the post-Helicobacter pylori era, its detection rate has been gradually increasing with the continuous improvement of endoscopic technology in China. Applying the PDCA cycle management in disease diagnosis can significantly improve the detection rate of the disease, benefiting patients. Through the PDCA management model, this study further enhanced gastroenterologists' understanding of this disease from various aspects, aiming to improve the clinical diagnosis of autoimmune gastritis.

ELIGIBILITY:
Inclusion Criteria:

Endoscopy center gastroenterologists in our hospital in 2024

Exclusion Criteria:

Doctors who withdrew from the PDCA management midway and stopped undergoing gastroscopy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Endoscopy center gastroenterologists in our hospital in 2024
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2024-08-15 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of AIG | 4months
  To diagnose Autoimmune Gastritis (AIG), the following two criteria must be simultaneously met:
  Endoscopic or histopathological findings, or both, that are consistent with the characteristics of autoimmune gastritis.
  Positive gastric autoantibody status, including the presence of anti-parietal cell antibodies (PCA) or anti-intrinsic factor antibodies (IFA), or both.
The suspected diagnosis rate of AIG | 4months
  If only the endoscopic or histopathological findings, or both, are consistent with the characteristics of autoimmune gastritis, but the gastric autoantibody status (anti-parietal cell antibodies or anti-intrinsic factor antibodies) is not confirmed to be positive, then the case should be considered as a suspected case of Autoimmune Gastritis (AIG).

SECONDARY OUTCOMES:
Parietal Cell Antibody（PCA） | 4months
  PCA is an important indicator in the diagnosis of AIG.
IF-Ab | 4months
  IFA is an important indicator in the diagnosis of AIG.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China